CLINICAL TRIAL: NCT05111379
Title: Acute Local Metabolomic Alterations in Blood and Muscle Tissue in Intermittent Claudication
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Tartu (Other)
Collaborators: Tartu University Hospital (Other); Estonian Science Foundation (Other Government)
Responsible Party: Principal Investigator, Jaak Kals, MD, Professor, University of Tartu
Other Study IDs: 350/T-2
Record Dates: First submitted 2021-09-28; First posted 2021-11-08 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Peripheral Arterial Occlusive Disease Fontaine Stage IIa
Keywords: lower extremity arterial disease; peripheral artery disease; intermittent claudication; local; metabolism; metabolomics; arteriovenous gradients; biomarkers; inflammation; ischemia-reperfusion injury
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Inflammation; Reperfusion Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, frozen tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LEAD (Fontaine IIa): Patients with mild intermittent claudication.
- Control: Healthy controls.

SUMMARY:
The most common clinical presentation of lower extremity arterial disease is intermittent claudication. Current understanding of the pathophysiology of intermittent claudication, as well as its treatment options are limited. The progression of the disease may lead to lower limb amputation, which is devastating for patients' quality of life and is a huge socio-economic burden to society.

Current study allows to determine the acute local metabolomic alterations in the ischaemic limb of the patient with intermittent claudication, and investigate the associations between the metabolomic alterations and the patient's maximal walking distance. This provides potentially valuable insight into the pathophysiology of this disease, and helps lay the groundwork for identifying potential novel targets for instituting more effective therapies for this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* LEAD group: Patients with diagnosis of lower extremity arterial disease (Fontaine IIa).
* Control group: Healthy volunteers with no leg symptoms and an ankle-brachial index (ABI) of 1.0-1.4.

Exclusion Criteria:

* Fontaine stages I or IIb-IV
* Exacerbation of limb ischaemia within the preceding 2 weeks;
* strong rest pain of any cause;
* age <18 or >80 years;
* fasting < 6 hours;
* time since last use of tobacco products < 6 hours;
* body mass index ≥ 35 kg/m2
* poor sonographic visibility of femoral artery;
* angina;
* cardiac arrhythmia at the time of presentation;
* presence of cardiac pacemaker;
* myocardial infarction within the preceding 3 months;
* stroke within the preceding 6 months;
* ongoing anticoagulant therapy;
* ongoing dual antiplatelet therapy;
* any revascularization within the preceding 3 month;
* marked heart failure (NYHA III-IV);
* blood pressure ≥ 180/110 mmHg;
* blood pressure <100/70 mmHg;
* clinically significant heart valve disease;
* acute infectious disease;
* active malignancy or chemotherapy or disease-free < 5 years;
* type I diabetes or insulin therapy;
* other clinically significant and untreated endocrine disorders;
* moderate to severe bronchial asthma (GINA 2016);
* severe chronic obstructive pulmonary disease (mMRC grade 3-4);
* acute (KDIGO 2012) or chronic renal disease (eGFR-EPI <30mL/min/1.73 m2);
* acute or chronic liver disease;
* anemia (<110 g/L);
* neuroinflammatory or neurodegenerative disease;
* active rheumatism;
* other diseases and factors that markedly hinder the subject's ability to walk during the treadmill exercise.
* For control group exclusively: history of lower extremity arterial disease / ABI <1.0 or >1.4.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with mild intermittent claudication (Fontaine IIa).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-01-28 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in local metabolomic profile after treadmill exercise as reflected by arteriovenous gradients of low-molecular metabolites. | Blood sampling at two points in time: Baseline (Day 1) & 10-15 minutes after treadmill test (Day 2).
  Measured using liquid chromatography combined with mass spectrometry (AbsoluteIDQ MxP Quant 500 Kit, BIOCRATES Life Sciences AG, Austria).
Change in local inflammatory profile after treadmill exercise as reflected by arteriovenous gradients of inflammatory mediators (IL-6, MPO, SOD, NOX isoform 1, NOX isoform 2, NOX isoform 5, nitrotyrosine, 8-iso-PGF2α). | Blood sampling at two points in time: Baseline (Day 1) & 10-15 minutes after treadmill test (Day 2).
  Measured using enzyme linked immunosorbent assay. Measurement unit: ng/mL.

SECONDARY OUTCOMES:
Change in local metabolomic profile after treadmill exercise as reflected by absolute concentrations of low-molecular metabolites in muscle biopsy. | Biopsy at two points in time: Baseline (Day 1) & 15-20 minutes after treadmill test (Day 2).
  Measured using liquid chromatography combined with mass spectrometry (AbsoluteIDQ MxP Quant 500 Kit, BIOCRATES Life Sciences AG, Austria).
Correlations between maximal walking distance and exercise-induced changes in local metabolomic and inflammatory profiles. | Data analysis after the enrollment period.
Correlations between baseline arterial functionality/hemodynamic parameters and exercise-induced changes in local metabolomic and inflammatory profiles. | Data analysis after the enrollment period.

OTHER OUTCOMES:
Maximal walking distance on a treadmill (m). | During treadmill test (Day 2).
Ankle-brachial index (no units). | Baseline (Day 1).
Femoral artery intima-media thickness (mm). | Baseline (Day 1).
Peripheral blood pressure, central blood pressure (mmHg). | Baseline (Day 1).
Aortic pulse wave velocity (m/s). | Baseline (Day 1).
Aortic augmentation index (%). | Baseline (Day 1).
Identification of systemic metabolomic profile as reflected by absolute concentrations of low-molecular metabolites in peripheral blood sample. | Blood sampling at one point in time: Baseline (Day 1)
  Measured using liquid chromatography combined with mass spectrometry (AbsoluteIDQ MxP Quant 500 Kit, BIOCRATES Life Sciences AG, Austria).
Identification of systemic inflammatory profile as reflected by absolute concentrations of inflammatory mediators (IL-6, MPO, SOD, NOX isoform 1, NOX isoform 2, NOX isoform 5, nitrotyrosine, 8-iso-PGF2α) in peripheral blood sample. | Blood sampling at one point in time: Baseline (Day 1)
  Measured using enzyme linked immunosorbent assay. Measurement unit: ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Jaak Kals, MD, PhD, Principal Investigator — University of Tartu; Kaido Paapstel, MD, PhD, Study Chair — University of Tartu; Kalle Kilk, MD, PhD, Study Chair — University of Tartu; Holger Post, MD, Study Chair — University of Tartu
Locations (1):
- Tartu University Hospital, Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Endothelial Research Centre — https://endothelialcentre.ut.ee/